CLINICAL TRIAL: NCT05303896
Title: Investigating Myocardial Remodelling in the Failing Human Heart
Acronym: RELAX
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ivar Sjaastad, Professor, Oslo University Hospital
Other Study IDs: 230524
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: MRI; Heart transplantation; Heart failure; PET
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Despite improvements in therapy, heart failure is a disease with high mortality and accelerating prevalence. To improve patient care, it is necessary to better understand the features and underlying mechanisms of myocardial remodeling; how it manifests in vivo and its underlying cellular and extracellular changes. The RELAX study will offer insight into myocardial remodeling, by comprehensively assessing function and structure of failing human hearts, and investigate its underlying cellular and extracellular changes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for heart transplantation
* Willingness to participate in the present study and ability to understand and sign the written informed consent

Exclusion Criteria:

* Patients under the age of 18.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients eligible for heart transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
MRI functional parameters including Left Ventricular Ejection Fraction and Global Longitudinal Strain | 1 years
  Measurement of myocardial function by in-vivo methods. In-vivo myocardial function will be obtained by MRI and echocardiography. Measurements include LVEF and GLS.
MRI morphological parameters including LVEDV and LVESV. | 1 years
  Measurement of myocardial morphology by in-vivo methods including MRI and ultrasound. The expected outcome in regards to morphology is varying degrees of geometrical abnormalities.
Myocardial stiffness measured by MRI and ex-vivo methods. | 1 year
  Measurement of myocardial stiffness by in-vivo and ex-vivo methods. In-vivo myocardial stiffness will be measured by MRI. The expected outcome is varying degrees of stiffness in accordance with the underlying pathology as well as regionally in the heart. Ex-vivo methods include stiffness measurements by histology and protein analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Sjaastad, MD, PhD, Principal Investigator — University of Oslo, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No